CLINICAL TRIAL: NCT02122510
Title: The Value of Preemptive Dexmedetomidine Transversus Abdominis Plane (TAP) Block in Patients Undergoing Elective Cesarean Section Under General Anesthesia.
Brief Title: Transverse Abdominal Block for Analgesia in Casarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ayman Abd Al-maksoud Yousef, Assistant Professor, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 1004/02/12
Record Dates: First submitted 2014-04-22; First posted 2014-04-24 (Estimated); Last update posted 2014-12-16 (Estimated); Status verified 2014-12

CONDITIONS: Analgesia Disorder
Keywords: Analgesia, casarean section, TAP block
MeSH Terms: conditions — Agnosia | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- dexmetomedine group (Active Comparator): dexmetomedine group will receive pre-delivery bilateral TAP block with 10 ml of bupivacaine 0.5 % mixed with 10 ml saline and 10 μg dexmetonedine in 20 ml syringe labeled G 2.
  Interventions: Drug: Dexmedetomidine
- Bupivacaine group (Active Comparator): Bupivacaine group will receive post-delivery bilateral TAP block with 10 ml of bupivacaine 0.5 % mixed with 10 ml saline in 20 ml syringe labeled G 2.
  Interventions: Drug: Bupivacine group

INTERVENTIONS:
Drug: Bupivacine group — Bupivacaine group(n=30) will receive post-delivery bilateral TAP block with 10 ml of bupivacaine 0.5 % mixed with 10 ml saline and 10 μg dexmetonedine in 20 ml syringe
  Other Names: Bucaine
  Arms: Bupivacaine group
Drug: Dexmedetomidine — Dexamedtomedine group will receive post-delivery bilateral TAP block with 10 ml of bupivacaine 0.5 % mixed with 10 ml saline and 10 μg dexmetonedine in 20 ml syringe
  Other Names: precdex
  Arms: dexmetomedine group

SUMMARY:
In this study, the investigators will compare the analgesic effect of bupivacaine and bupivacaine-dexmetomedine after elective cesarean delivery by performing an bilateral TAP block, on the patients for whom the operation will be performed under general anesthesia.

DETAILED DESCRIPTION:
The investigators will study 60 ASA [American Society of Anesthesiologist] physical status I and ІІ patients undergoing elective cesarean delivery at tanta University Hospital, in a prospective, randomized, comparative, clinical trial.

Patients will be randomly allocated to two equal groups (n = 30) using closed envelopes labeled 1,and 2 reflecting group 1and 2 respectively.

The drugs are prepared by the anesthesiologist who is not involved in the study or data collection.

Group I: (n=30) will receive pre-delivery bilateral TAP block with 10 ml of bupivacaine 0.5 % mixed with 10 ml saline and 10 μg dexmetonedine in 20 ml syringe labeled G 2.

Group II: (n=30) will receive post-delivery bilateral TAP block with 10 ml of bupivacaine 0.5 % mixed with 10 ml saline in 20 ml syringe labeled G2.

ELIGIBILITY:
Inclusion Criteria:

1. We will study 60 ASA [American Society of Anesthesiologist] physical status I and ІІ patients undergoing elective cesarean delivery
2. Age between 21-40 years old.

Exclusion Criteria:

1. Refusal of participation in the study
2. Patients who have infection or tumor at the site of puncture for local anesthetic injection.
3. Patients who have coagulopathy, platelet abnormalities, and concurrent treatment with anticoagulant drugs.
4. Patients known to have allergy or sensitivity to dexmetomedine, and/or bupivacaine
5. Severe hepatic and/or renal insufficiency
6. Morbid obesity (body mass index (BMI) >35)
7. Psychological disease

Ages: 21 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2013-03; Primary Completion 2014-05 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
hemodynamic changes | 2 hours
  blood pressure and heart rate measured every 15 minutes during the intraopertive peroid

SECONDARY OUTCOMES:
Analgesic requirements | 24 hours
  VAS will be measured during 24 hours after surgery every 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Ayman A Yousef, MD, Principal Investigator — Assistant professor; Ayman A Yousef, MD, Study Director — Assistant Professor
Locations (1):
- Tanta University Hospitals, Tanta, Algharbiya, Egypt